CLINICAL TRIAL: NCT05105672
Title: A Single-Arm, Single-Center Phase II Clinical Study of Sintilimab Combined With Concurrent Chemoradiation Therapy in The Treatment of Stage IIA2 To IVA (2018 FIGO) Locally Advanced Cervical Cancer
Brief Title: A Study of Sintilimab Combined With Concurrent Chemoradiation Therapy in Locally Advanced Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI308XZH
Record Dates: First submitted 2021-10-25; First posted 2021-11-03 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Uterine Cervical Neoplasms; Sintilimab
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — sintilimab; Cisplatin; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chemoradiotherapy + Sintilimab (Experimental): Participants will be given intravenous administration of sintilimab (200mg, q3w), cisplatin(75 mg/m², q3w) and Radiotherapy. After completing 2 cycles of concurrent chemoradiation, the Participants will continue to use 4 cycles of sintilimab (200mg, q3w) and cisplatin(75 mg/m², q3w) as maintenance therapy.
  Interventions: Drug: Sintilimab; Drug: Cisplatin; Radiation: External Beam Radiotherapy (EBRT); Radiation: brachytherapy

INTERVENTIONS:
Drug: Sintilimab — IV infusion
Drug: Cisplatin — IV infusion
Radiation: External Beam Radiotherapy (EBRT) — Undergo pelvic EBRT
Radiation: brachytherapy — brachytherapy

SUMMARY:
This is a single-arm, single-center phase II clinical study to explore the efficacy and safety of sintilimab combined with concurrent chemoradiation therapy as treatment in women with locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Has high-risk locally advanced cervical cancer (LACC): The International Federation of Gynecology and Obstetrics (FIGO) 2018 Stage IB3 or FIGO 2018 Stages IIA2-IVA.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Has radiographically evaluable disease, either measurable or non-measurable per RECIST 1.1
* Adequate hematological, renal and hepatic functions:Hemoglobin > 9.0 g/dl; Neutrophils > 2000 cells/μl; ANC > 1.5 × 10^9/L;Platelets > 100 × 10^9/L;

Exclusion Criteria:

* Has received prior therapy with an anti-programmed cell death receptor 1 (PD-1), anti-programmed cell death receptor ligand 1 (PD-L1), or anti-programmed cell death receptor ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX-40, CD137).
* Has a known history of Human Immunodeficiency Virus (HIV) infection.
* Prior malignancies (other than curable non-melanoma skin cancer) within 5 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 1 year
  The proportion of patients with at least one tumor scan of complete response (CR) or partial response (PR) using RECIST v1.1

SECONDARY OUTCOMES:
Progression free survival | Time from diagnosis of disease to disease progression or death due to any cause
  2 years
Overall survival | Time from diagnosis of disease of treatment until death due to any cause
  2 years
Incidence of ADRs and tolerance | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Longzhen Zhang, MD, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China